CLINICAL TRIAL: NCT03991013
Title: AntiRetroviral Therapy In Second-line: Investigating Tenofovir-lamivudine-dolutegravir (ARTIST): a Randomised Controlled Trial
Brief Title: Tenofovir-lamivudine-dolutegravir Combination as Second-line ART: a Randomised Controlled Trial
Acronym: ARTIST
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Cape Town (Other)
Collaborators: Wellcome Trust (Other); Médecins Sans Frontières, Belgium (Other)
Responsible Party: Principal Investigator, Graeme Meintjes, Professor of Medicine, University of Cape Town (UCT), University of Cape Town
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ARTIST
Record Dates: First submitted 2019-05-31; First posted 2019-06-19 (Actual); Results first posted 2024-08-09 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: HIV Infections
Keywords: second line antiretroviral therapy; dolutegravir
MeSH Terms: conditions — HIV Infections | interventions — dolutegravir

STUDY DESIGN:
Intervention Model Description: This study will be a phase 2, randomised, double-blind, placebo-controlled trial of tenofovir-lamivudine-dolutegravir fixed-dose combination daily with a lead-in supplementary 50 mg dose of dolutegravir versus matching placebo taken 12 hours later for the first 14 days in patients failing a first-line tenofovir-emtricitabine/lamivudine-efavirenz regimen.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Supplementary dose (Active Comparator): Tenofovir-lamivudine-dolutegravir fixed-dose combination tablet daily with an additional dolutegravir 50 mg dose taken 12 hours later for the first 14 days.
  Interventions: Drug: Dolutegravir 50 mg
- Placebo dose (Placebo Comparator): Tenofovir-lamivudine-dolutegravir fixed-dose combination tablet daily with a matching placebo taken 12 hours later for the first 14 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dolutegravir 50 mg — Tenofovir-lamivudine-dolutegravir fixed-dose combination tablet with a lead-in supplementary dose of 50 mg dolutegravir taken 12 hours later for the first 14 days, with continuation of tenofovir-lamivudine-dolutegravir for the duration of the study (48 weeks).
  Other Names: Dalimune 50 mg
  Arms: Supplementary dose
Drug: Placebo — Tenofovir-lamivudine-dolutegravir fixed-dose combination tablet with a matching placebo taken 12 hours later for the first 14 days, with continuation of tenofovir-lamivudine-dolutegravir for the duration of the study (48 weeks).
  Arms: Placebo dose

SUMMARY:
The strategy to support virological suppression on second-line antiretroviral treatment (ART) includes the provision of ART that has a low pill burden, good tolerability, low toxicity, is easily monitored, has a high barrier to resistance, and that is low cost. The fixed-dose combination of tenofovir-lamivudine-dolutegravir offers significant advantage as a potential second-line regimen compared to the World Health Organization standard of care second-line regimen of zidovudine-lamivudine-dolutegravir, in terms of cost, tolerability and monitoring requirements.

The ARTIST study is a phase 2, randomised, double-blind, placebo-controlled trial aiming to determine the proportion of patients achieving virological suppression when recycling the tenofovir-emtricitabine/lamivudine backbone with dolutegravir (tenofovir-lamivudine-dolutegravir fixed-dose combination) as a second-line with and without a lead-in supplementary dose of dolutegravir, in patients failing a tenofovir-emtricitabine/lamivudine-efavirenz first-line regimen.

There is evidence to suggest that even in the presence of resistance mutations to tenofovir and lamivudine (K65R or M184V/I), using this backbone with dolutegravir will provide an effective second-line regimen in patients who have failed a first-line regimen of tenofovir-emtricitabine/lamivudine-efavirenz. The strategy of giving a lead-in supplementary dose of dolutegravir is in view of the inducing effect of efavirenz on dolutegravir metabolism and transport that persists for 2 weeks after efavirenz is stopped; the inducing effect decreases with time after efavirenz is stopped.

Given that these patients will have elevated viral loads, a high baseline risk of nucleoside reverse transcriptase inhibitor (NRTI) resistance and efavirenz resistance, and the inducing effect of efavirenz on dolutegravir metabolism and transport that persists for 2 weeks, this study will comprise two stages. The first stage will evaluate virological suppression in 62 participants initiated on the fixed-dose combination of tenofovir-lamivudine-dolutegravir with a lead-in supplementary dose of dolutegravir for the first 14 days. The study will progress to the second stage if this strategy proves effective, and 130 participants will then be randomised to receive the fixed-dose combination of tenofovir-lamivudine-dolutegravir with and without this lead-in dose.

The primary endpoint is virological suppression (viral load <50 copies/mL) at 24 weeks.

A pharmacokinetic sub-study will be conducted on 12 participants in stage 1 and 24 participants in stage 2, to assess the trough concentrations of dolutegravir and off-treatment concentrations of efavirenz at day 3, 7, 14, and 28. This is to evaluate the need for the lead-in supplementary dose of dolutegravir.

ELIGIBILITY:
Inclusion Criteria:

HIV positive patients over 18 years old, who have failed first-line ART regimen of tenofovir-emtricitabine/lamivudine-efavirenz, are able to attend the study clinic for one year of scheduled visits and who have given written, informed consent will be enrolled in this study. In female patients of child-bearing potential, those willing to use effective and reliable contraception for the duration of the study will be eligible.

Failure of a first-line regimen is defined as a viral load (VL) of >1000 copies/mL (within the previous two months) and an immediately prior VL >1000 copies/mL, taken 2-24 months prior (based on data captured by National Health Laboratory Service).

Exclusion Criteria:

* If the patient has two VLs 2-3 months apart: >2 log drop in VLs between the most recent VL (within the previous two months) and the immediately prior VL (taken 2-3 months prior)
* CD4 count <100 cells/microlitre
* Estimated glomerular filtration rate (eGFR) <50 mL/min/1.73 m2 using the Modification of Diet in Renal Disease (MDRD) formula
* Alanine aminotransferase >100 U/L or total bilirubin >twice the upper limit of normal
* Pregnant or desire to become pregnant during the study period (48 weeks)
* Breastfeeding
* Being treated for active tuberculosis (TB) or concern that patient has undiagnosed active TB (based on symptom screening) as rifampicin reduces the concentrations of dolutegravir and thus requires dose adjustments
* Any current diagnosis of malignancy
* Allergy or intolerance to one of the drugs in regimen
* Active, severe psychiatric disease judged likely to impact adherence
* Current substance abuse judged likely to impact adherence
* On treatment for AIDS-defining condition (not including secondary prophylaxis maintenance therapy)
* Any other clinical condition that in the opinion of an investigator puts the patient at increased risk if participating in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 192 (Actual)
Dates: Start 2019-08-08 (Actual); Primary Completion 2022-04-26 (Actual); Study Completion 2022-10-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Graeme Meintjes, PhD, Principal Investigator — University of Cape Town; Claire Keene, Principal Investigator — Médecins Sans Frontières, Belgium
Locations (1):
- Khayelitsha Site B/Ubuntu Community Health Clinic, Cape Town, Western Cape, South Africa

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared with other organisations or individuals for further research upon a reasonable request to the University of Cape Town PI, provided that certain conditions are met (including but not limited to the ethical standards upheld by Human Research Ethics Committee (HREC) that approved the initial study).
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: From the time the final results are published
Access Criteria: Data will be shared with other organisations or individuals for further research upon a reasonable request to the University of Cape Town PI, provided that certain conditions are met (including but not limited to the ethical standards upheld by HREC that approved the initial study).

REFERENCES:
- [Derived] Griesel R, Banda CG, Zhao Y, Omar Z, Wiesner L, Meintjes G, Sinxadi P, Maartens G. Pharmacokinetics of Single-Dose Versus Double-Dose Dolutegravir After Switching From a Failing Efavirenz-Based Regimen. J Acquir Immune Defic Syndr. 2024 May 1;96(1):85-91. doi: 10.1097/QAI.0000000000003402. PMID 38372621
- [Derived] Keene CM, Cassidy T, Zhao Y, Griesel R, Jackson A, Sayed K, Omar Z, Hill A, Ngwenya O, Van Zyl G, Flowers T, Goemaere E, Maartens G, Meintjes G. Recycling Tenofovir in Second-line Antiretroviral Treatment With Dolutegravir: Outcomes and Viral Load Trajectories to 72 weeks. J Acquir Immune Defic Syndr. 2023 Apr 15;92(5):422-429. doi: 10.1097/QAI.0000000000003157. PMID 36706364
- [Derived] Zhao Y, Griesel R, Omar Z, Simmons B, Hill A, van Zyl G, Keene C, Maartens G, Meintjes G. Initial Supplementary Dose of Dolutegravir in Second-Line Antiretroviral Therapy: A Noncomparative, Double-Blind, Randomized Placebo-Controlled Trial. Clin Infect Dis. 2023 May 24;76(10):1832-1840. doi: 10.1093/cid/ciad023. PMID 36645792
- [Derived] Zhao Y, Keene C, Griesel R, Sayed K, Gcwabe Z, Jackson A, Ngwenya O, Schutz C, Goliath R, Cassidy T, Goemaere E, Hill A, Maartens G, Meintjes G. AntiRetroviral Therapy In Second-line: investigating Tenofovir-lamivudine-dolutegravir (ARTIST): protocol for a randomised controlled trial. Wellcome Open Res. 2021 Feb 17;6:33. doi: 10.12688/wellcomeopenres.16597.1. eCollection 2021. PMID 36017341

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Stage 1 of the ARTIST study was a single-arm prospective cohort study of second-line TLD regimen with supplementary dolutegravir dose (50 mg twice daily) for two weeks in patients failing a NNRTI-based regimen. After completion of stage 1, the study progressed to enrol 130 participants in stage 2.
Groups:
- Stage 2: Supplementary Dose; Stage 1: TLD Regimen With Supplementary Dolutegravir Dose: Tenofovir-lamivudine-dolutegravir fixed-dose combination tablet daily with an additional dolutegravir 50 mg dose taken 12 hours later for the first 14 days.
  Dolutegravir 50 mg: Tenofovir-lamivudine-dolutegravir fixed-dose combination tablet with a lead-in supplementary dose of 50 mg dolutegravir taken 12 hours later for the first 14 days, with continuation of tenofovir-lamivudine-dolutegravir for the duration of the study (48 weeks).
- Stage 2: Placebo Dose: Tenofovir-lamivudine-dolutegravir fixed-dose combination tablet daily with a matching placebo taken 12 hours later for the first 14 days.
  Placebo: Tenofovir-lamivudine-dolutegravir fixed-dose combination tablet with a matching placebo taken 12 hours later for the first 14 days, with continuation of tenofovir-lamivudine-dolutegravir for the duration of the study (48 weeks).
Period: Overall Study
Arm/Group | Stage 2: Supplementary Dose | Stage 2: Placebo Dose | Stage 1: TLD Regimen With Supplementary Dolutegravir Dose
Started | 65 | 65 | 62
Completed | 64 | 63 | 62
Not Completed | 1 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Stage 2: Supplementary Dose | Stage 2: Placebo Dose | Stage 1: TLD Regimen With Supplementary Dolutegravir Dose | Total
Number analyzed (Participants) | 65 | 65 | 62 | 192
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 38 [33 to 45] | 39 [34 to 45] | 37 [31 to 46] | 38 [32 to 45]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42 | 47 | 43 | 132
  Male | 23 | 18 | 19 | 60
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black | 65 | 65 | 62 | 192
Weight [Median (Inter-Quartile Range); unit: kg] | 74 [62 to 87] | 80 [63 to 96] | 71 [62 to 81] | 77 [62 to 88]
BMI [Median (Inter-Quartile Range); unit: kg/m2] | 28.4 [23.1 to 33.8] | 30.1 [24.4 to 35.5] | 27.8 [22.6 to 32.4] | 29.0 [23.5 to 35.1]
CD4 cell count [Median (Inter-Quartile Range); unit: cells/μL] | 246 [187 to 334] | 250 [154 to 349] | 259 [175 to 380] | 246 [160 to 337]
HIV-1 RNA [Median (Inter-Quartile Range); unit: log10 copies/mL] | 4.12 [3.46 to 4.69] | 4.01 [3.51 to 4.66] | 3.98 [3.45 to 4.57] | 4.02 [3.48 to 4.68]
Time receiving first-line ART [Median (Inter-Quartile Range); unit: months] | 77 [45 to 112] | 93 [57 to 132] | 62 [34 to 98] | 88 [51 to 119]
Two fully active NRTIs [Count of Participants; unit: Participants] — Population: Denominators indicate the numbers of participants with available viral sequences.
  Participants
    number analyzed (Participants) | 63 | 57 | 56 | 176
    (all) | 2 | 2 | 6 | 10
Resistance to 1 NRTI [Count of Participants; unit: Participants] — Population: Denominators indicate the numbers of participants with available viral sequences
  Participants
    number analyzed (Participants) | 63 | 57 | 56 | 176
    (all) | 15 | 10 | 14 | 39
Resistance to both NRTIs [Count of Participants; unit: Participants] — Population: Denominators indicate the numbers of participants with available viral sequences
  Participants
    number analyzed (Participants) | 63 | 57 | 56 | 176
    (all) | 46 | 45 | 36 | 127
TFV-DP concentration [Median (Inter-Quartile Range); unit: fmol/punch] | 948 [725 to 1253] | 1052 [733 to 1437] | 1186 [859 to 1905] | 960 [729 to 1388]

OUTCOME MEASURES:

1. Primary Outcome: Virological Suppression at 24 Weeks
Description: Proportion of participants with HIV viral load <50 copies/mL at 24 weeks analysed by modified intention to treat (ITT) and according to the FDA snapshot algorithm
Time Frame: 24 weeks
Population: mITT analysis excludes those switching study drug for reasons of stopping contraception or desire to become pregnant, becoming pregnant, transfer out for nonclinical reasons, and death from non-HIV and nondrug causes.
Measure: Count of Participants; unit: Participants
Arm/Group | Stage 2: Supplementary Dose | Stage 2: Placebo Dose | Stage 1: TLD Regimen With Supplementary Dolutegravir Dose
Number analyzed (Participants) | 64 | 65 | 62
Participants | 55 | 53 | 53

2. Secondary Outcome: Virological Suppression at 24 Weeks (Sensitivity Analysis)
Description: Proportion of participants with HIV viral load <50 copies/mL at 24 weeks using pre-specified sensitivity analyses
Time Frame: 24 weeks
Population: Sensitivity analysis excludes those excluded from mITT analysis, as well as loss to follow-up, missing viral load within the window, switching study drug for reasons other than treatment failure, and evidence of poor adherence (tenofovir diphosphate <350 fmol/punch).
Measure: Count of Participants; unit: Participants
Arm/Group | Stage 2: Supplementary Dose | Stage 2: Placebo Dose | Stage 1: TLD Regimen With Supplementary Dolutegravir Dose
Number analyzed (Participants) | 64 | 61 | 60
Participants | 55 | 53 | 53

3. Secondary Outcome: Virological Suppression at 12 Weeks (Modified ITT)
Description: Proportion of participants with HIV viral load <50 copies/mL at 12 weeks analysed by modified ITT.
Time Frame: 12 weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Stage 2: Supplementary Dose | Stage 2: Placebo Dose | Stage 1: TLD Regimen With Supplementary Dolutegravir Dose
Number analyzed (Participants) | 64 | 65 | 60
Participants | 53 | 55 | 45

4. Secondary Outcome: Antiretroviral Resistance Mutations by Genotypic Resistance Testing
Description: To describe dolutegravir resistance or emergent resistance mutations to tenofovir or lamivudine in participants eligible for genotypic resistance testing by 24 weeks
Time Frame: 24 weeks
Population: If any HIV-1 RNA after week 12 was ≥50 copies/mL, or if there was <1 log10 decline in HIV-1 RNA from baseline, or if HIV-1 RNA was suppressed and sub- sequently rebound to ≥50 copies/mL, enhanced adherence counseling was performed, and HIV-1 RNA measurement was repeated after 2 weeks. If the repeat HIV-1 RNA was ≥500 copies/mL, a genotypic antiretroviral resistance test was performed.
Measure: Count of Participants; unit: Participants
Arm/Group | Stage 2: Supplementary Dose | Stage 2: Placebo Dose | Stage 1: TLD Regimen With Supplementary Dolutegravir Dose
Number analyzed (Participants) | 3 | 3 | 1
Participants | 0 | 0 | 0

5. Secondary Outcome: CD4 Change at 24 Weeks
Description: Change in CD4 count from screening to week 24
Time Frame: 24 weeks
Measure: Median (Inter-Quartile Range); unit: cells/μL
Arm/Group | Stage 2: Supplementary Dose | Stage 2: Placebo Dose | Stage 1: TLD Regimen With Supplementary Dolutegravir Dose
Number analyzed (Participants) | 65 | 65 | 62
cells/μL | 88 [45 to 138] | 75 [18 to 127] | 99 [36 to 163]

6. Secondary Outcome: Adverse Events
Description: To describe grade 3 or 4 adverse events and serious adverse events
Time Frame: 24 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Stage 2: Supplementary Dose | Stage 2: Placebo Dose | Stage 1: TLD Regimen With Supplementary Dolutegravir Dose
Number analyzed (Participants) | 65 | 65 | 62
Participants | 4 | 5 | 12

7. Secondary Outcome: All-cause Mortality
Description: To describe all-cause mortality.
Time Frame: 24 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Stage 2: Supplementary Dose | Stage 2: Placebo Dose | Stage 1: TLD Regimen With Supplementary Dolutegravir Dose
Number analyzed (Participants) | 65 | 65 | 62
Participants | 1 | 0 | 0

8. Secondary Outcome: Adherence to Treatment
Description: To describe tenofovir-diphosphate (TFV-DP) concentrations (ng/mL) at 24 weeks
Time Frame: 24 weeks
Population: We monitored adherence with tenofovir diphosphate (TFV-DP) concentrations using stored dried blood spot specimens.
Measure: Median (Inter-Quartile Range); unit: fmol/punch
Arm/Group | Stage 2: Supplementary Dose | Stage 2: Placebo Dose | Stage 1: TLD Regimen With Supplementary Dolutegravir Dose
Number analyzed (Participants) | 63 | 64 | 62
fmol/punch | 1354 [930 to 1873] | 1393 [1098 to 1811] | 1186 [859 to 1905]

9. Secondary Outcome: Geometric Mean Ratio (GMR) of Dolutegravir Trough Concentrations on Day 7 Versus Day 28
Description: To evaluate the geometric mean ratio (GMR) of dolutegravir trough concentrations on day 7 versus day 28
Time Frame: First 28 days
Measure: Geometric Mean (90% Confidence Interval); unit: ratio
Arm/Group | Stage 2: Supplementary Dose | Stage 2: Placebo Dose | Stage 1: TLD Regimen With Supplementary Dolutegravir Dose
Number analyzed (Participants) | 13 | 11 | 12
ratio | 1.654 [1.404 to 1.948] | 0.637 [0.485 to 0.837] | 1.654 [1.404 to 1.948]

ADVERSE EVENTS:
Time Frame: 48 weeks
Description: Adverse events were evaluated and graded at all study visits according to the Division of AIDS Table for Grading the Severity of Adult and Paediatric Adverse Events.
Arm/Group | Stage 2: Supplementary Dose | Stage 2: Placebo Dose | Stage 1: TLD Regimen With Supplementary Dolutegravir Dose
All-Cause Mortality (participants affected / at risk) | 1/65 | 0/65 | 0/62
Serious Adverse Events (participants affected / at risk) | 2/65 | 0/65 | 9/62
Other Adverse Events (participants affected / at risk) | 2/65 | 5/65 | 3/62
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Stage 2: Supplementary Dose (N=65) | Stage 2: Placebo Dose (N=65) | Stage 1: TLD Regimen With Supplementary Dolutegravir Dose (N=62)
severe COVID-19 (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
acute psychosis (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
fractured tibia (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
urinary tract infection (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
incident pulmonary tuberculosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
stab chest (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
perianal abscess (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
condylomata acuminata (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Stage 2: Supplementary Dose (N=65) | Stage 2: Placebo Dose (N=65) | Stage 1: TLD Regimen With Supplementary Dolutegravir Dose (N=62)
acute psychosis (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
incident pulmonary tuberculosis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
raised random glucose (Endocrine disorders) | 0 (0) | 2 (2) | 0 (0)
acute kidney injury (Renal and urinary disorders) | 0 (0) | 2 (2) | 1 (1)
headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
raised blood pressure (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2020-06-17): https://cdn.clinicaltrials.gov/large-docs/13/NCT03991013/Prot_005.pdf
  • Statistical Analysis Plan (2022-05-09): https://cdn.clinicaltrials.gov/large-docs/13/NCT03991013/SAP_007.pdf
  • Informed Consent Form (2020-06-17): https://cdn.clinicaltrials.gov/large-docs/13/NCT03991013/ICF_006.pdf